CLINICAL TRIAL: NCT05793372
Title: Hyperhomocysteinemia in Alzheimer's Disease
Acronym: Hcy-MA
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENAUD Mathilde, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI049
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease; Homocystinemia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Alzheimer's Disease: Patients with Alzheimer's disease
  Interventions: Other: Retrospective study of clinical features

INTERVENTIONS:
Other: Retrospective study of clinical features — Retrospective study of clinical features

SUMMARY:
Alzheimer's disease (AD) is the most common neurodegenerative disease. Age is its main risk factor. AD is a multifactorial disease, combining genetic and environmental risk factors. Autosomal dominant mutations have been identified (PSEN1, PSEN2, APP), leading to earlier and more severe forms of the disease. Other genetic risk factors have been identified, such as the ε4 allele of the APOE gene. . The environment also plays a major role, with the identification of several risk factors such as air pollution or nutritional deficiencies.

AD patients frequently present hyperhomocysteinemia, a consequence of a dysfunction of monocarbon metabolism. Homocysteine is an amino acid involved in the metabolism of methionine and cysteine. High concentrations of homocysteine can be deleterious to the central nervous system.

Most prospective studies have shown that elevated homocysteine is a predictor of undefined cognitive impairment or AD. Other studies have focused on clinical data and, in particular, on cognitive function. For example, a meta-analysis found an inverse correlation between MMSE score and homocysteine level.

Thus, our study seeks to evaluate the impact of hyperhomocysteinemia on the severity and early onset of AD, while knowing the presence or absence of genetic risk factors associated with AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease
* Positive CSF biomarkers
* age of onset < 75 years
* already benefited from a previous research of Alzheimer's disease genetic features (PSEN1, PSEN2, APP, APOE)
* already benefited from a previous research of homocysteine cycle (monocarbon metabolism) by complete exome/clinical exome or panel

Exclusion Criteria:

* patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's disease with positive CSF biomarkers, age of onset < 75 years, and having already benefited from a previous research of Alzheimer's disease genetic features (PSEN1, PSEN2, APP, APOE) and homocysteine cycle (monocarbon metabolism) by complete exome/clinical exome or panel
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between homocysteine levels and the severity/early onset of Alzheimer's disease | baseline
  Mesure of homocysteine levels Mesure of MiniMental State Evaluation (MMSE), age of symptoms onset

SECONDARY OUTCOMES:
Evaluation of the frequency of hyperhomocysteinemia in a homogeneous population of patients with Alzheimer's disease. | baseline
  measurement of homocysteine levels in our cohort (µmol/L)
Evaluation of the genetic characteristics of Alzheimer's disease Evaluation of the genetic characteristics of homocysteine monocarbon metabolism. | baseline
  search for an autosomal dominant mutation (APP, PSEN1 or PSEN2) or a risk factor mutation for Alzheimer's disease (TREM2, SORL1, ABCA7) and APOE status search for a mutation in the genes of monocarbon metabolism
Evaluation of the frequency of vitamin B deficiencies in a homogeneous population of patients with Alzheimer's disease. | baseline
  measurement of B1,B6,B9 and B12 levels in our cohort (nmol/L)